CLINICAL TRIAL: NCT03045237
Title: Sporty Bellies - Intervention Program During Pregnancy on Women and Newborn
Brief Title: Healthy Bellies - Intervention Program During Pregnancy on Women and Newborn
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Minho (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other); Centro de Investigação em Estudos da Criança (Unknown); Centro Hospitalar do Alto Ave (Unknown); Câmara Municipal de Guimarães (Unknown)
Responsible Party: Principal Investigator, Ana Isabel Teixeira Jesus Silva, PhD Student, University of Minho
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Healthy Bellies
Record Dates: First submitted 2017-01-28; First posted 2017-02-07 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Lifestyle; Physical Activity; Dietary Habits; Depressive Symptoms
Keywords: Pregnancy; Physical activity; Newborn; Depressive Symptoms; Dietary habits; Healthy lifestyles
MeSH Terms: conditions — Motor Activity; Feeding Behavior; Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The program consists in 3 physical exercise classes, one of them in the pool.
  Interventions: Other: physical exercises classes
- Control Group (No Intervention): The control group has the basic information through health professionals.

INTERVENTIONS:
Other: physical exercises classes — 3 physical exercises classes, one of them in the pool.
  Arms: Intervention Group

SUMMARY:
"Healthy Bellies" is an intervention program with pregnant women, based on the promotion of healthy lifestyles. It aims to evaluate the impact of the program in the health of both pregnant and newborn. This trial is being conducted with pregnant women, divided into control and intervention group. Are performed 3 assessment periods: 1 - beginning of the program; 2 - postpartum; 3 - 1 month after delivery. The intervention group has a program of 3 weekly physical exercise classes and the control group has the basic information that is usually provided by health professionals. With this program, it is expected to contribute with evidence to the best practice in the field of interventions in pregnancy and improve health outcomes of both pregnant and newborn.

ELIGIBILITY:
Inclusion Criteria:

* Do not have any medical or obstetric contraindication for physical exercise

Exclusion Criteria:

* Haemodynamically significant heart disease;
* restrictive lung disease;
* incompetent cervix/cerclage;
* multiple gestation at risk for premature labor;
* persistent second or third trimester bleeding;
* placenta praevia after 26 weeks gestation;
* premature labor during the current pregnancy;
* ruptured membranes;
* pregnancy induced hypertension;
* severe anaemia;
* unevaluated maternal cardiac arrhythmia;
* chronic bronchitis;
* poorly controlled type I diabetes;
* extreme morbid obesity;
* extreme underweight (body mass index <12);
* history of extremely sedentary lifestyle;
* intrauterine growth restriction in current pregnancy;
* poorly controlled hypertension/pre-eclampsia;
* orthopaedic limitations;
* poorly controlled seizure disorder;
* poorly controlled thyroid disease; heavy smoker).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in physical activity assessed with the "Pregnancy Physical Activity Questionnaire" | Baseline and 1 month after delivery
  Evaluation through "Pregnancy Physical Activity Questionnaire"
Change in Dietary intake assessed with the "Food frequency questionnaire" | Baseline and 1 month after delivery
  Evaluation through "Food frequency questionnaire"
Gestational Weight gain | 1 day after delivery
  Values are self-reported by pregnant women
Change in Depressive Symptoms assessed with the "Edinburgh Postnatal Depression Scale" | Baseline, 1 day after delivery and 1 month after delivery
  Evaluation through "Edinburgh Postnatal Depression Scale"
Weight of the baby | 1 day after delivery
  Self-reported by participants
Length of the baby | 1 day after delivery
  Self-reported by participants

CONTACTS AND LOCATIONS:
Overall Officials: Maria B Pereira, Study Director — University of Minho
Locations (1):
- Universidade do Minho, Braga, Portugal

IPD SHARING:
Plan to Share IPD: Undecided